CLINICAL TRIAL: NCT04454203
Title: Femoral Peri-arterial Local Anesthetic Injection Via Peri-arterial Perineural Catheter Reverses Tourniquet Associated Ischemic Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00104144
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Tourniquet Hypertension; Intraoperative Hypertension; Total Ankle Arthroplasty; Ankle Fusion
Keywords: Perifemoral; Tourniquet; Mepivacaine; Tourniquet Hypertension
MeSH Terms: interventions — Mepivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepivacaine Block Group (Experimental): Infiltration of local anesthetic (mepivacaine) above and beside the femoral artery through a perineural catheter.
  Interventions: Drug: Mepivacaine; Procedure: Perifemoral Injection of Local Anesthetic
- Saline Sham Group (Placebo Comparator): Infiltration of salt water (saline) above and beside the femoral artery through a perineural catheter.
  Interventions: Drug: Saline; Procedure: Perifemoral Injection of Local Anesthetic

INTERVENTIONS:
Drug: Mepivacaine — An infiltration of mepivacaine superomedially to the femoral artery via perineural catheter.
  Other Names: Carbocaine
  Arms: Mepivacaine Block Group
Drug: Saline — An infiltration of saline superomedially to the femoral artery via perineural catheter.
  Other Names: Salt water placebo
  Arms: Saline Sham Group
Procedure: Perifemoral Injection of Local Anesthetic — Infiltration of mepivacaine superomedially to the formal artery via perineural catheter in an effort to numb the nerves that contribute to tourniquet hypertension intraoperatively.
  Other Names: Femoral Periarterial Injection
  Arms: Mepivacaine Block Group
Procedure: Perifemoral Injection of Local Anesthetic — Infiltration of saline superomedially to the formal artery via perineural catheter that should NOT numb the nerves that contribute to tourniquet hypertension intraoperatively.
  Other Names: Femoral Periarterial Injection
  Arms: Saline Sham Group

SUMMARY:
The goal of this prospective randomized double-blind study is to determine if an ultrasound guided peri-arterial injection of local anesthetic (LA) superomedially the femoral artery via peripheral nerve catheter reverses ischemic hypertension associated with prolonged lower extremity tourniquet time.

DETAILED DESCRIPTION:
This is a research study to find out if injection of numbing medication by the large artery going down your leg will improve high blood pressure caused by the tourniquet.

Depending on whether you enroll in this study, you may receive an injection of local anesthetic (numbing medication) or saline (salt water) by your femoral artery (the large artery going down your leg). This is to see how this injection impacts your blood pressure during surgery as the surgeons use a tourniquet (device that squeezes your leg) to help decrease the bleeding during surgery. Oftentimes the tourniquet causes your blood pressure to go up, but the numbing medication may help return your blood pressure close to its normal level. The rest of your anesthesia care, including other nerve blocks and general anesthetic, will be the same as it would be without participating in the study. You will be enrolled in this study for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

Patients that will be included in the study are English speaking 18-75 year old ASA 1-3 patients undergoing total ankle arthroplasty.

Exclusion Criteria:

1. ASA 4 or 5
2. Diagnosis of chronic pain
3. Daily chronic opioid use (over 3 months of continuous opioid use).
4. Inability to communicate pain scores or need for analgesia.
5. Infection at the site of block placement
6. Age under 18 years old or greater than 75 years old
7. Pregnant women (as determined by standard of care day-of surgery urine bHCG)
8. Intolerance/allergy to local anesthetics
9. Weight <50 kg
10. Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
11. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance.
12. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Change in tourniquet hypertension as measured by systolic blood pressure | From time of injection to 30 minutes after injection
  Infiltrating study drug to reverse intraoperative tourniquet hypertension

SECONDARY OUTCOMES:
Pain Scores (NRS11) | Perioperative start until 2 hours after admission to PACU
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Opioid consumption | Perioperative start until 2 hours after admission to PACU
  Perioperative opioid consumption as measured in oral morphine equivalents (OMEs)
Quadriceps motor function | 1 hour after extubation
  Gross quadriceps motor function as measured by leg extension

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kumar, MD, PhD, Principal Investigator — Duke University; William M Bullock, MD, PhD, Study Director — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; patients will be deidentified and no personal information or medical records used.